CLINICAL TRIAL: NCT04599452
Title: Safety and Efficacy of Allogeneic NK Cell Therapy for Recurrent/Refractory Elderly AML
Brief Title: NK Cell Therapy Recurrent/Refractory Elderly AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020NKAML
Record Dates: First submitted 2020-09-11; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: AML; Recurrent; Refractory; Elderly
Keywords: Recurrent/Refractory Elderly AML NK cell
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 patients with recurrent refractory elderly AML were treated (Experimental): The aim of this investigation was to assess safety and efficacy of allogenic NK cells therapy for recurrent refractory elderly AML.
  Interventions: Biological: Allogeneic NK cell regimen group

INTERVENTIONS:
Biological: Allogeneic NK cell regimen group — 10 patients with recurrent refractory elderly AML were treated with allogeneic NK cell regimen.
  Allogeneic NK cell regimen ×3 cycle; Cyclophosphamide 300mg/m2.d d1to 3; G-CSF 150ug bid d4-11; Azacitidine 75mg/m2 d5-11; Allogeneic NK cell 10-30×10^6/kg d13，d15.

SUMMARY:
The aim of this investigation was to assess safety and efficacy of allogenic NK cells therapy for recurrent refractory elderly AML.

ELIGIBILITY:
Inclusion Criteria:

1. The 2 or more than 2-cycles of standard regimen was used to treat elderly AML patients who did not achieve complete remission or relapse.
2. Patients with age 60 years to 70 years.
3. KPS greater than or equal to 60.
4. ALT and AST are less than 3 times normal.
5. Total bilirubin less than 1.5mg/dl(25.65umol/L).
6. Serum creatinine less than 2.5mg/dl(221umol/L), or creatinine scavenging ability greater than or equal to 60 mL/min/1.73 m2.
7. Left ventricular ejection fraction cardiac greater than or equal to 45%, Echocardiography (ECHO) showed no pericardial effusion, Electrocardiogram (ECG) is normal.
8. No pleural effusion in lungs
9. Oxyhemoglobin saturation greater than or equal to 92% in normal environment.
10. KIR mismatch between patient and umbilical cord blood.
11. Volunteer to participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Malignant tumor patient.
2. Patients who are accompanied by fungal, bacterial, viral, or other uncontrolled infections or require level 4 isolation( HBV-DNA quantification and normal liver function in patients with hepatitis b infection are excluded).
3. Patients with HIV, HCV positive.
4. Patients with central nervous system diseases, including stroke, epilepsy, dementia, or autoimmune central nervous system disorders.
5. During the first 12 months of enrollment, patients with cardioangiography or stents, active angina pectoris or other clinically significant symptoms, or with cardiogenic asthma.
6. Patients receiving anticoagulant therapy or with severe coagulation disorders.
7. According to the researcher's judgment, the drug treatment the patient is receiving will affect the safety and effectiveness of the study.
8. Patients with allergies or history of allergies to biological agents used in this program.
9. Systemic steroid used within 2 weeks before treatment (except for recent or present use of inhaled corticosteroids).
10. Patients with other uncontrolled diseases, Investigators think it is not suitable for the participants.
11. Any circumstance that the investigator considers may increase the risk to the subject or interfere with the results of the study.
12. Patients participate in other clinical studies.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (PR+CR) | 3 months
  The proportion of patients with complete response(CR) or partial response(PR) as measured by response criteria definitions for acute myeloid leukemia

SECONDARY OUTCOMES:
Overall survival(OS) | 1 year
  The proportion of patients with overall survival(OS).

CONTACTS AND LOCATIONS:
Overall Officials: Chengyun Zheng, Ph.D., Study Director — The Second Hospital of Shandong University
Locations (1):
- The 2nd Hospital of Shandong University, Jinan, Shandong, China